CLINICAL TRIAL: NCT06059157
Title: Epileptogenic Network Visualisation With Advanced MRI
Acronym: EPIVAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/26JUI/281
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Drug Resistant Epilepsy
Keywords: epilepsy; network; non-invasive investigation
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single Arm
  Interventions: Device: Advanced MRI

INTERVENTIONS:
Device: Advanced MRI — resting-state functional MRI, diffusion with advanced post-processing (microstructure analysis), myelin mapping

SUMMARY:
The goal of this clinical trial is to improve non-invasive identification of epileptogenic networks in drug-resistant epileptic patient.

The investigators aim to compare epileptogenic network identification with stereo-EEG (used as glod standard) with the identification of the same network using advanced MRI (rs-fMRI, microstructural analysis of white matter, ...). The main goals are to:

1. Compare the accuracy of network identification.
2. Analyse the effect of the MRI sequences on candidates selection and target identification.

Participants will already have been selected for stereoEEG and will undergo a supplementary MRI (about 1h) with the additional MRI sequences. Follow-up MRI are scheduled for patient undergoing a second, therapeutic epileptic surgery.

DETAILED DESCRIPTION:
Patient identified for SEEG will undergo, prior to the implantation procedure an MRI with the following sequences:

* 3D T1
* rsfMRI
* multishell diffusion

The rsfMRI will be post-processed to delineate the epileptogenic networks based on an Independant Component Analysis (ICA) methods. Once the epileptogenic network(s) has/have been identified, connexion between the different regions will be identified through post-processing of the diffusion using a MSMT-CSD algorithm. Finally, the identified tract between the different region will be quantitatively analysed using different algorithms (NODDI, DIAMOND, MF) to better grasp there integrity.

In a follow-up study, the patients that will later on benefit from a resection or disconnection (i.e. curative surgery) will also have an identical MRI 3 months after the said procedure to evaluate the evolution on the network(s) based on the same criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from drug-resistant epilepsy
* Patient already selected for SEEG implantation as part of their epileptic networks

Exclusion Criteria:

* Patient excluded from SEEG (pregnant women, children too young for the procedure, patient unable to undergo the procedure)
* Contra-indication for MRI

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Network identification with MRI | At the end of phase 1 - expected to be 3 years after first inclusion
  Analysis of the anatomical overlap of radiological network (with MRI) and the electrophysiological network (with SEEG) using coregistration and a sublobar analysis. Overlap will be quantified in %.
Prognosis of network targetting with surgery | One year after surgery (phase 2)
  Analysis of the impact on epileptic outcome in accordance with effect of the surgery on the network. The impact of the surgery on the network will be assessed by coregistration to determine which part of the network has been removed or disconnected. The epileptic outcome will be assessed using the Engel classification
Interest of adding epileptic network radiological analysis in a standard epileptic work-up | Approximately 1 year after the start of phase 3
  Analyse the impact on therapeutic and/or diagnostic decision of the network radiological analysis in a standard clinical practice. This impact will be assessed by measuring the change in the type of decision (further work-up, invasive EEG, "curative" surgery, "palliative" surgery or no modification) or the modification in the extent of surgery (more/less electrodes for invasive EEG, more/less tissue targeted with surgery)

SECONDARY OUTCOMES:
Network quantification | At the end of phase 1 - expected to be 3 years after first inclusion
  Analysis of the strength of the network using radiological data (r², Z-score, diffusion metrics obtained via microfingerprinting such as fiber volume fraction and fiber fraction) vs electrophysiological metrics (epileptogenic index, h²)
Network regulation with surgery | One year after surgery (phase 2)
  Analysis of the impact of the surgery on the radiological parameters of the network cited in outcome 4 (r² and Z-score for rsfMRI, number of tracts for tractography and strenght of tract with fiber fraction and fiber volume fraction for microfingerprinting)

CONTACTS AND LOCATIONS:
Overall Officials: Riëm El Tahry, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires St-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be kept on RedCap and made available after reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after completion of the study
Access Criteria: reasonable request evaluated by the research team